CLINICAL TRIAL: NCT01244685
Title: Randomized Controlled Trial With Deltex CardioQ in Elective Bowel Resection Patients
Brief Title: Trial With Deltex Cardio in Elective Bowel Resection Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Roberto Bergamaschi, Professor and Chief, Division of Colon and Rectal Surgery, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 139939
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: 1 Fluid Management
Keywords: bowel resection; Deltex CardioQ Probe; fluid management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- probe (Active Comparator): Patients in the 'goal-directed fluid' Lactated Ringers solution according to ideal body weight for the first 24 hours. The fluids will be changed after the first 24 hours and continued until the patient is tolerating a regular diet. The Deltex CardioQ esophageal probe will be evaluated every 15 minutes in the Post Anesthesia Care Unit (PACU) by the Anesthesia service. Stroke Volume (SV), Flow Time Corrected (FTc), and Peak Velocity (PV) will be measured. A short FTc (<330 ms) indicative of hypovolemia will receive a 3cc/kg fluid challenge with Lactated Ringers crystalloid solution over 5 minutes. A SV increase of >10% will receive a further 3cc/kg fluid challenge. A SV increase of <10% will not receive further fluid challenge.
  Interventions: Device: Deltex CardioQ Probe
- Standard Fluid (No Intervention): Patients in the 'standard fluid' group will receive Lactated Ringers solution for 24 hours post-operatively at 1 times maintenance rate according to ideal body weight. Then the fluids will be changed to physiologic maintenance with D5½NS at the same rate. Fluids will be decreased by ½ once the patient is tolerating a clear liquid diet, and then discontinued once the patient is tolerating a regular diet.

INTERVENTIONS:
Device: Deltex CardioQ Probe — Deltex CardioQ probe will be placed nasally in the operating room by the anesthesia team and fluid management will be administered via anesthesia protocol.
  Arms: probe

SUMMARY:
The purpose of this study is:

* To determine if the intraoperative fluid administration with the Deltex CardioQ esophageal Doppler will reduce the length of stay after elective bowel resection.
* The probe can be used to dynamically measure stroke volume and cardiac output. This information will assist us in determining the ideal amount of fluids to be administered.
* To determine if the fluid administration established by the esophageal probe will result in a shorter length of stay in elective bowel resection patients.
* The investigators plan to enroll 100 patients in this study.

DETAILED DESCRIPTION:
Intraoperative goal-directed IV fluid administration utilizing an esophageal Doppler as a guide to measuring the amount of fluid by looking into the stroke volume to determine if there is too little or too much fluid. It has been shown that inadequate fluid administration is a cause of increased morbidity and length of stay after elective bowel resection. However, there are no data evaluating the Doppler's use in the postoperative period, only intraoperatively. Our objective is to evaluate whether postoperative goal-directed fluid management with the Deltex CardioQ esophageal Doppler probe leads to shorter hospital stay in elective bowel resection patients. All consecutive patients randomized into the 'standard fluid' group and the 'goal-directed fluid' group. All will follow standard surgical postoperative care with the exception of fluid administration. If eligible, all patients will receive an epidural catheter for pain control. The 'goal-directed fluid' group will have a Deltex CardioQ probe placed nasally in the operating room by the anesthesia team, and fluid management will be administered via anesthesia protocol. The 'standard fluid' group will not receive the Deltex CardioQ probe.Patients in the 'goal-directed fluid' group will receive fluids according to body weight for the first 24 hours. The probe will be evaluated every15 minutes in the Post Anesthesia Care Unit and measurements will be taken to determine whether fluids will be given to the patient.On the surgical floor, patients in the 'goal-directed fluid' group will be evaluated every 8 hours and fluids will be given if necessary according to measurements taken via the probe.

Intraoperative goal-directed IV fluid administration utilizing an esophageal Doppler as a guide to measuring the amount of fluid by looking into the stroke volume to determine if there is too little or too much fluid. It has been shown that inadequate fluid administration is a cause of increased morbidity and length of stay after elective bowel resection. However, there are no data evaluating the Doppler's use in the postoperative period, only intraoperatively. Our objective is to evaluate whether postoperative goal-directed fluid management with the Deltex CardioQ esophageal Doppler probe leads to shorter hospital stay in elective bowel resection patients. All consecutive patients randomized into the 'standard fluid' group and the 'goal-directed fluid' group. All will follow standard surgical postoperative care with the exception of fluid administration. If eligible, all patients will receive an epidural catheter for pain control. The 'goal-directed fluid' group will have a Deltex CardioQ probe placed nasally in the operating room by the anesthesia team, and fluid management will be administered via anesthesia protocol. The 'standard fluid' group will not receive the Deltex CardioQ probe.Patients in the 'goal-directed fluid' group will receive fluids according to body weight for the first 24 hours. The probe will be evaluated every15 minutes in the Post Anesthesia Care Unit and measurements will be taken to determine whether fluids will be given to the patient.On the surgical floor, patients in the 'goal-directed fluid' group will be evaluated every 8 hours and fluids will be given if necessary according to measurements taken via the probe.

ELIGIBILITY:
Inclusion Criteria:

* All elective bowel resection cases, laparoscopic or open
* Age 18 or older
* Ability to consent

Exclusion Criteria:

* All emergency cases
* Inability to consent
* Esophageal or upper airway disease or recent surgery
* Moderate or severe aortic valvular disease, congestive heart failure
* Severe kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Length of stay | at Discharge
  Length of hospital stay from day of admission to day of discharge

SECONDARY OUTCOMES:
Determining the ideal amount of fluids to be administered | During and post surgery
  • The probe can be used to dynamically measure stroke volume and cardiac output. This information will assist us in determining the ideal amount of fluids to be administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Broook University Medical Center, Stony Brook, New York, United States